CLINICAL TRIAL: NCT06457282
Title: Studying The Association Between Environmental Exposure to Polyfluoroalkyl Substances and Breast Cancer in Assiut Governorate- Egypt
Brief Title: Studying The Association Between Environmental Exposure to PFAS and Breast Cancer in Assiut Governorate- Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jacklin Farouk Danial Beshay, Demonstrator, Assiut University
Other Study IDs: Breast Cancer andPFAS exposure
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case ( breast cancer patients)
- Control ( Healthy people without breast cancer)

SUMMARY:
1. Measuring serum level of PFAS in breast cancer female patients and healthy participants.
2. Studying the correlation between serum level of PFAS and breast cancer risk through statistical modeling and analysis.
3. Studying the magnitude of environmental exposure through measuring levels of PFAS in air and water sources of corresponding participants.

DETAILED DESCRIPTION:
* Perfluoroalkyl substances (PFASs) are persistent pollutants that are present in the environment.
* Perfluorooctanoic acid (PFOA) and perfluorooctane sulfonate (PFOS), known as the most detected per- and polyfluoroalkyl substances (PFAS)in various environmental compartments.They have been associated with plastic pollution and endocrine dysfunction.

Humans are exposed to PFASs through various pathways, including dietary items such as seafood, drinking water, and some dental floss.. Contaminated drinking water and food supply are potential sources of 0ral exposure to PFAS PFASs have been used in various products such as firefighting foams, surfactants, non-stick pans, food contact materials such as boxes, bags, wrappers, cups, (Lim, 2019), and table wares, and personal care products including cosmetics.

Over the past 180 years (1839-2019), numerous emerging contaminants have been identified, Perfluorooctanoic acid (PFOA) and perfluoro octane sulfonate (PFOS) are two of the most used PFAS compounds in various applications and have already been identified as endocrine-disrupting chemicals(EDCs).

Due to their structural and functional similarities with endogenous steroid hormones, EDCs mimic and interfere with homeostatic mechanisms and signaling pathways of hormones in the body even at low concentrations. They cause a variety of endocrine and metabolic disorders ,developmental abnormalities and hormone-dependent cancers.

PFAS exhibits a wide range of toxic effects, including developmental toxicity, genotoxicity, carcinogenicity, hepatotoxicity, reproductive toxicity, immunotoxicity, cytotoxicity, neurotoxicity, and hormonal toxicity.

Moreover, the International Agency for Research on Cancer (IARC) has classified PFOA as "possibly carcinogenic to humans".

Breast cancer is one of the major female health problems worldwide. Although there is growing evidence indicating that pollution increases the risk of breast cancer, there is still inconsistency among previous studies.

As we mentioned before, that PFAS is considered as EDC.so it may interact with estrogen receptors (ATSDR, 2018). And multiple studies found association between PFOS exposure and decreasd serum or saliva concentrations of estrogen in women.

It is well known that breast cancer is hormone-dependent, its development may be associated with exposure to xenoestrogens found in environmental pollutants (Adami et al., 2018).

Multiple epidemiological (Morgan et al., 2017) and experimental studies (Pierozan et al., 2018; Pierozan and Karlsson, 2018;) have associated EDC exposure with increased risk of breast cancer and breast cancer metastasis.Exposure to some PFASs has been both positively (Mancini et al., 2020; Tsai et al., 2020) associated with breast cancer risk as in Greenlandic Inuit women.and inversely associated with breast cancer risk as inTaiwanese women.

The presented study will be the first study to be done in Egypt to study the risk of PFAS environmental exposure and its correlation to breast cancer. Currently, there is no information available on the production, use, management and bio persistence of PFAS substances in Egypt. This is an area that needs attention, particularly for substances dispersed directly into the environment such as PFAS. And performing a risk assessment study identifying high exposure levels to various PFAS compounds in Assiut Governorate which will help in establishing the PFAS Egyptian toxicological report recommended by the Ministry of Environment as a part of the Stockholm Convention to protect human health and the environment from persistent organic pollutants.With increasing concerns of climate changes and global warming Egypt proceeded in setting recommendations for PFAS elimination.These recommendation contributes to the achievement of several key Sustainable Development Goals (SDGs) due to the impacts of the substances on health and ecosystems including water pollution.

ELIGIBILITY:
Inclusion Criteria:

-

Newly diagnosed cases. Who are diagnosed by ultrasonography and mammography and confirmed diagnosis after biopsy taken for histopathological examination.

Exclusion Criteria:

* 1. Patients who underwent neoadjuvant chemotherapy prior to their surgery will be excluded from the study.

  2.To eliminate confounding factors, breast cancer patients with comorbidities and chronic diseases such as uncontrolled diabetes mellitus or other endocrine disorders, poorly controlled hypertension, acute coronary syndrome, congestive heart failure, chronic kidney disease and chronic liver disease will be excluded.

  3.Women with biopsy-proven benign breast disease should be excluded

  .4. Patients who have other malignancies are excluded

  6. patients with family history of breast cancer will be excluded. 7. Patients refuse to continue the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female women age group between 18: 65 years. 2. Newly diagnosed cases. Who are diagnosed by ultrasonography and mammography and confirmed diagnosis after biopsy taken for histopathological examination
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
1- Measuring serum level of PFAS in breast cancer female patients and healthy participants. | 2 yrs
  Studying the correlation between serum level of PFAS and breast cancer risk through statistical modeling and analysis.
  Studying the magnitude of environmental exposure through measuring levels of PFAS in air and water sources of corresponding participants.

REFERENCES:
- [Background] Tsai MS, Chang SH, Kuo WH, Kuo CH, Li SY, Wang MY, Chang DY, Lu YS, Huang CS, Cheng AL, Lin CH, Chen PC. A case-control study of perfluoroalkyl substances and the risk of breast cancer in Taiwanese women. Environ Int. 2020 Sep;142:105850. doi: 10.1016/j.envint.2020.105850. Epub 2020 Jun 21. PMID 32580117
- [Background] Itoh H, Harada KH, Kasuga Y, Yokoyama S, Onuma H, Nishimura H, Kusama R, Yokoyama K, Zhu J, Harada Sassa M, Tsugane S, Iwasaki M. Serum perfluoroalkyl substances and breast cancer risk in Japanese women: A case-control study. Sci Total Environ. 2021 Dec 15;800:149316. doi: 10.1016/j.scitotenv.2021.149316. Epub 2021 Jul 29. PMID 34392213
- [Background] Pierozan P, Cattani D, Karlsson O. Tumorigenic activity of alternative per- and polyfluoroalkyl substances (PFAS): Mechanistic in vitro studies. Sci Total Environ. 2022 Feb 20;808:151945. doi: 10.1016/j.scitotenv.2021.151945. Epub 2021 Nov 27. PMID 34843762
- [Background] Velarde MC, Chan AFO, Sajo MEJV, Zakharevich I, Melamed J, Uy GLB, Teves JMY, Corachea AJM, Valparaiso AP, Macalindong SS, Cabaluna ND, Dofitas RB, Giudice LC, Gerona RR. Elevated levels of perfluoroalkyl substances in breast cancer patients within the Greater Manila Area. Chemosphere. 2022 Jan;286(Pt 1):131545. doi: 10.1016/j.chemosphere.2021.131545. Epub 2021 Jul 12. PMID 34293563